CLINICAL TRIAL: NCT04233255
Title: The Role of Neuromuscular Ultrasound in Diagnosis of Muscle Diseases
Brief Title: Role of Ultrasound in Diagnosis of Muscle Diseases
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manar Nasr Abd-el-hakim Nasr, principal investigator, Assiut University
Other Study IDs: RUDM
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Ultrasound; Muscle Disease
Keywords: Ultrasound; Muscle; Electrophysiology
MeSH Terms: conditions — Muscular Diseases | interventions — Electrophysiologic Techniques, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with muscle disease(myositis, hereditary myopathy): Includes 64 symptomatic patients with muscle disease subdivided into two subgroups (a) 10 patients with acute inflammatory myositis; And (b 545patients with hereditary myopathy. The patients will be subjected to neuromuscular ultrasound (US) and electrophysiology at baseline,after 6 months and after 12 months. The number and location of studied muscles will be determined according to pattern of clinical presentation.
  Interventions: Device: Neuromuscular Ultrasound (US); Device: Electrophysiological studies; Diagnostic Test: Seum CPK, CK-MM levels, Lactate dehydrogenase and alanine aminotransferase.
- Healthy volunteers as control group: Includes 64 healthy volunteers as control group. They will be subjected to neuromuscular ultrasound (US) and electrophysiology at baseline. Their age, sex, number and location of studied muscles will be matched with patients' group.
  Interventions: Device: Neuromuscular Ultrasound (US); Device: Electrophysiological studies; Diagnostic Test: Seum CPK, CK-MM levels, Lactate dehydrogenase and alanine aminotransferase.

INTERVENTIONS:
Device: Neuromuscular Ultrasound (US) — Quantitative ultrasound measurements will be performed to studied muscles according to a standard protocol; for each muscle three consecutive measurements will be made to minimize variation in echo intensity during analysis .The captured images will be analyzed offline for echo intensity by means of computer-assisted grayscale histogram analysis.The study will be performed using My lab 7 ultrasound system (Esaote company, Italy) that is equipped by 7-19 MHz linear array transducer and color and power Doppler.
  Technique: evaluation of studied muscles for echo intensity (ECHO), quantitative assessments of echointensity, muscle perfusion, transverse and longitudinal sections of the muscle and its thickness at rest and during maximal voluntary contractions (MVC), overlying subcutaneous fat, cross-sectional area (CSA), and angled fibers of pennate muscles.
Device: Electrophysiological studies — Includes: Motor and sensory nerve conduction study, F-wave and H-reflex study to assess the proximal roots, Electromyography (EMG) of the studied muscles.
  using machine: recordings will be performed with a Nihon Kohden equipment (model 7102) with the following parameters: sweep time 8 ms/D, sensitivity 0.5 mV/D, low frequency filter 2 Hz, high frequency filter 10 kHz, stimulation duration 0.1 ms and stimulation frequency 1 Hz.
Diagnostic Test: Seum CPK, CK-MM levels, Lactate dehydrogenase and alanine aminotransferase. — measured in U/L using ELISA.

SUMMARY:
The study aims to provide a timely update on the role of combining clinical and neuromuscular ultrasound assessments in diagnosis and follow-up of various muscle diseases in clinical practice over 12 months period, and correlating US findings with functional scales, biochemical and electrophysiological studies.

DETAILED DESCRIPTION:
Many muscle diseases share common clinical features that render arriving at appropriate diagnoses difficult. The combination of muscle imaging with clinical can limit the differential diagnosis and yield the most probable one and can direct genetic testing as the only method to arrive at a definite diagnosis.

In recent years, the use of high-resolution ultrasound had become an important tool in diagnosis and in the monitoring of disease progression and treatment of both hereditary and acquired myopathies. Additionally, it entails a safe, accessible, low-cost, and no ionizing radiation tool which renders the technique extremely suitable for paediatric patients and patients who cannot lie still without sedation. therefore, it can be used as a complementary tool to electro-diagnosis.

Ultrasound permits to evaluate echo intensity, muscle perfusion, transverse and longitudinal sections of the muscle and its thickness at rest and during maximal voluntary contractions, overlying subcutaneous fat, cross-sectional area, and angled fibers of pennate muscles.

The use of sonographically guided biopsy is an easy, safe, and reliable method for attaining tissue for histologic diagnosis in neuromuscular disease.

In most myopathies, either acute or chronic, muscle tissue undergoes morphological changes giving rise to replacement of muscle by connective tissue and/or fat. Pattern recognition on muscle imaging might be helpful in distinguishing between different disease entities.

ELIGIBILITY:
Inclusion Criteria:

* Males and females.
* 2-60 years old.
* For patients with acute inflammatory myositis: patients presenting with characteristic picture of acute inflammatory myositis according to the myositis association 2019.
* For patients with acute inflammatory myositis: newly diagnosed patients within one month from onset of disease.
* All patients not received any previous specific treatment for myopathy.

Exclusion Criteria:

* Patients with clinically or electrophysiologically suspected other neuromuscular conditions that mimic myopathy such as motor neuron disease, neuromuscular junction disorders.
* Patients with secondary causes of myopathies; as drug induced, endocrinal disorders like diabetes mellitus and hypothyroidism or metabolic myopathy.
* Patients who received any previous specific treatment for myopathy

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will be performed on 2 groups Group (I): 32 patients diagnosed to have muscle disease subdivided into two subgroups (a)16 patients with acute inflammatory myositis; And (b)16 patients with hereditary myopathy. Group (II): including 32 healthy volunteers matching age and sex as control group.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
The rate of decline of patients with muscle disorder versus normal subjects as assessed by quantitative ultrasound measurements and electrophysiology studies. | up to 12 months
  With the successful completion of this aim, the investigators will establish that alterations in both quantitative ultrasound and electromyography will provide meaningful measures of disease progression.

SECONDARY OUTCOMES:
Rate of change in Functional assessment of muscle weakness | up to 12 months
  Grading score from 0-10 according to affected muscles
Rate of change in manual muscle strength testing by EXPANDED MRC (The modified Medical Research Council) | up to 12 months
  Grading scale from 0 -5 points, measures strength of each muscle group score 0 is the weakest (worst) and 5 is the strongest (best)
Rate of change of serum CPK and CK-MM levels | up to 12 months
  measured in U/L using ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Nageh F. El-Gammal, Doctorate, Study Chair — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wattjes MP, Kley RA, Fischer D. Neuromuscular imaging in inherited muscle diseases. Eur Radiol. 2010 Oct;20(10):2447-60. doi: 10.1007/s00330-010-1799-2. Epub 2010 Apr 27. PMID 20422195
- [Result] Boon A. Ultrasonography and electrodiagnosis: are they complementary techniques? PM R. 2013 May;5(5 Suppl):S100-6. doi: 10.1016/j.pmrj.2013.03.014. Epub 2013 Mar 19. PMID 23524068
- [Result] Chiaramonte R, Bonfiglio M, Castorina EG, Antoci SAM. The primacy of ultrasound in the assessment of muscle architecture: precision, accuracy, reliability of ultrasonography. Physiatrist, radiologist, general internist, and family practitioner's experiences. Rev Assoc Med Bras (1992). 2019 Feb;65(2):165-170. doi: 10.1590/1806-9282.65.2.165. PMID 30892439
- [Result] O'Sullivan PJ, Gorman GM, Hardiman OM, Farrell MJ, Logan PM. Sonographically guided percutaneous muscle biopsy in diagnosis of neuromuscular disease: a useful alternative to open surgical biopsy. J Ultrasound Med. 2006 Jan;25(1):1-6. doi: 10.7863/jum.2006.25.1.1. PMID 16371549
- [Result] Kubinova K, Dejthevaporn R, Mann H, Machado PM, Vencovsky J. The role of imaging in evaluating patients with idiopathic inflammatory myopathies. Clin Exp Rheumatol. 2018 Sep-Oct;36 Suppl 114(5):74-81. Epub 2018 Oct 1. PMID 30296982
- [Result] Mah JK, van Alfen N. Neuromuscular Ultrasound: Clinical Applications and Diagnostic Values. Can J Neurol Sci. 2018 Nov;45(6):605-619. doi: 10.1017/cjn.2018.314. PMID 30430964
- [Result] Barohn RJ, Dimachkie MM, Jackson CE. A pattern recognition approach to patients with a suspected myopathy. Neurol Clin. 2014 Aug;32(3):569-93, vii. doi: 10.1016/j.ncl.2014.04.008. PMID 25037080
- [Result] Vanhoutte EK, Faber CG, van Nes SI, Jacobs BC, van Doorn PA, van Koningsveld R, Cornblath DR, van der Kooi AJ, Cats EA, van den Berg LH, Notermans NC, van der Pol WL, Hermans MC, van der Beek NA, Gorson KC, Eurelings M, Engelsman J, Boot H, Meijer RJ, Lauria G, Tennant A, Merkies IS; PeriNomS Study Group. Modifying the Medical Research Council grading system through Rasch analyses. Brain. 2012 May;135(Pt 5):1639-49. doi: 10.1093/brain/awr318. Epub 2011 Dec 20. PMID 22189568
- See also: Diagnostic criteria for inflammatory myositis — https://www.myositis.org/about-myositis/diagnosis/diagnostic-criteria/diagnostic-criteria-for-polymyositis/